CLINICAL TRIAL: NCT02087514
Title: Duration of Red Blood Cell Storage Prior to Transfusion and Non-Transferrin-Bound Iron
Brief Title: Duration of Red Blood Cell Storage Prior to Transfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven L. Spitalnik, Professor of Pathology and Cell Biology, Columbia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: AAAI0835; R01HL115557 (NIH)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Iron, Blood Level Abnormal
Keywords: Blood Transfusion; Iron; Red Blood Cells
MeSH Terms: interventions — Blood Transfusion; Erythrocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Transfusion of PRBC stored for 1 week (Active Comparator): Subjects will receive blood transfusion with packed red blood cells stored for 1 week.
  Interventions: Procedure: Blood Transfusion; Other: Packed red blood cells
- Transfusion of PRBC stored for 2 weeks (Experimental): Subjects will receive blood transfusion with packed red blood cells stored for 2 weeks.
  Interventions: Procedure: Blood Transfusion; Other: Packed red blood cells
- Transfusion of PRBC stored for 3 weeks (Experimental): Subjects will receive blood transfusion with packed red blood cells stored for 3 weeks.
  Interventions: Procedure: Blood Transfusion; Other: Packed red blood cells
- Transfusion of PRBC stored for 4 weeks (Experimental): Subjects will receive blood transfusion with packed red blood cells stored for 4 weeks.
  Interventions: Procedure: Blood Transfusion; Other: Packed red blood cells
- Transfusion of PRBC stored for 5 weeks (Experimental): Subjects will receive blood transfusion with packed red blood cells stored for 5 weeks.
  Interventions: Procedure: Blood Transfusion; Other: Packed red blood cells
- Transfusion of PRBC stored for 6 weeks (Experimental): Subjects will receive blood transfusion with packed red blood cells stored for 6 weeks.
  Interventions: Procedure: Blood Transfusion; Other: Packed red blood cells

INTERVENTIONS:
Procedure: Blood Transfusion — A routine medical procedure in which blood is given through an intravenous (IV) line a blood vessel.
  Other Names: Red blood cell (RBC) transfusion
Other: Packed red blood cells — Red blood cells that have been collected, processed, and stored in bags as blood product units available for blood transfusion.
  A standard autologous leukoreduced packed red blood cell unit will be collected and stored in AS-3 solution in the Columbia University Medical Center blood bank.
  The number of weeks in storage are as follows:
  * 1 week
  * 2 weeks
  * 3 weeks
  * 4 weeks
  * 5 weeks
  * 6 weeks
  Other Names: PRBC

SUMMARY:
This study will determine the minimal duration of red blood cell (RBC) storage that leads to increases in circulating non-transferrin-bound iron in healthy human volunteers post-transfusion. The results from this study will help guide national guidelines for appropriate duration of RBC storage prior to transfusion, which is currently 6 weeks by Food and Drug Administration (FDA) criteria. The overall objective of this research is to improve the safety of refrigerated storage of red blood cells before transfusion.

DETAILED DESCRIPTION:
Recent studies suggest that older stored blood is associated with worse outcomes in certain hospitalized patients. Red cells may be stored in a refrigerator prior to transfusion for up to 42 days by current FDA standards. Refrigerator storage of red cells is associated with a storage lesion and the survival of transfused red cells decreases with increasing storage time, thus older blood is associated with an increased delivery of hemoglobin-iron to certain parts of the body. The investigators have preliminary data in mice and humans suggesting that delivery of a significant iron load from aged red cells leads to the production of a potentially toxic form of circulating iron called non-transferrin-bound iron.

In this prospective study of healthy volunteers, each subject will be randomized to receive transfusion of one RBC unit after 1, 2, 3, 4, 5, or 6 weeks of storage. The primary outcome will be the 24 hr area under the curve (AUC) of the serum non-transferrin bound iron concentration calculated from samples collected at 0, 2, 4, 6, 8, 10, 12, 14 and 24 hours after transfusion.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Body weight >110 lbs
* Hemoglobin >12.5 g/dL

Exclusion Criteria:

* Ineligible for donation based on the New York Blood Center blood donor questionnaire
* Systolic blood pressure >180 or <90 mm Hg, diastolic blood pressure >100 or <50 mm Hg
* Heart rate <50 or >100
* Temperature >99.5 F prior to donation
* Temperature >100.4 F or subjective feeling of illness prior to transfusion (this is to avoid having a concurrent illness affect post-transfusion measurements);
* Positive results on standard blood donor infectious disease testing
* Positive urine pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Spitalnik, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rapido F, Brittenham GM, Bandyopadhyay S, La Carpia F, L'Acqua C, McMahon DJ, Rebbaa A, Wojczyk BS, Netterwald J, Wang H, Schwartz J, Eisenberger A, Soffing M, Yeh R, Divgi C, Ginzburg YZ, Shaz BH, Sheth S, Francis RO, Spitalnik SL, Hod EA. Prolonged red cell storage before transfusion increases extravascular hemolysis. J Clin Invest. 2017 Jan 3;127(1):375-382. doi: 10.1172/JCI90837. Epub 2016 Dec 12. PMID 27941245

RESULTS

PARTICIPANT FLOW:
Groups:
- Transfusion of PRBC Stored for 1 Week: Subjects will receive blood transfusion with packed red blood cells stored for 1 week.
  Blood Transfusion: A routine medical procedure in which blood is given through an intravenous (IV) line a blood vessel.
  Packed red blood cells: Red blood cells that have been collected, processed, and stored in bags as blood product units available for blood transfusion.
  A standard autologous leukoreduced packed red blood cell unit will be collected and stored in AS-3 solution in the Columbia University Medical Center blood bank.
  The number of weeks in storage are as follows:
  * 1 week
  * 2 weeks
  * 3 weeks
  * 4 weeks
  * 5 weeks
  * 6 weeks
- Transfusion of PRBC Stored for 2 Weeks: Subjects will receive blood transfusion with packed red blood cells stored for 2 weeks.
  Blood Transfusion: A routine medical procedure in which blood is given through an intravenous (IV) line a blood vessel.
  Packed red blood cells: Red blood cells that have been collected, processed, and stored in bags as blood product units available for blood transfusion.
  A standard autologous leukoreduced packed red blood cell unit will be collected and stored in AS-3 solution in the Columbia University Medical Center blood bank.
  The number of weeks in storage are as follows:
  * 1 week
  * 2 weeks
  * 3 weeks
  * 4 weeks
  * 5 weeks
  * 6 weeks
- Transfusion of PRBC Stored for 3 Weeks: Subjects will receive blood transfusion with packed red blood cells stored for 3 weeks.
  Blood Transfusion: A routine medical procedure in which blood is given through an intravenous (IV) line a blood vessel.
  Packed red blood cells: Red blood cells that have been collected, processed, and stored in bags as blood product units available for blood transfusion.
  A standard autologous leukoreduced packed red blood cell unit will be collected and stored in AS-3 solution in the Columbia University Medical Center blood bank.
  The number of weeks in storage are as follows:
  * 1 week
  * 2 weeks
  * 3 weeks
  * 4 weeks
  * 5 weeks
  * 6 weeks
- Transfusion of PRBC Stored for 4 Weeks: Subjects will receive blood transfusion with packed red blood cells stored for 4 weeks.
  Blood Transfusion: A routine medical procedure in which blood is given through an intravenous (IV) line a blood vessel.
  Packed red blood cells: Red blood cells that have been collected, processed, and stored in bags as blood product units available for blood transfusion.
  A standard autologous leukoreduced packed red blood cell unit will be collected and stored in AS-3 solution in the Columbia University Medical Center blood bank.
  The number of weeks in storage are as follows:
  * 1 week
  * 2 weeks
  * 3 weeks
  * 4 weeks
  * 5 weeks
  * 6 weeks
- Transfusion of PRBC Stored for 5 Weeks: Subjects will receive blood transfusion with packed red blood cells stored for 5 weeks.
  Blood Transfusion: A routine medical procedure in which blood is given through an intravenous (IV) line a blood vessel.
  Packed red blood cells: Red blood cells that have been collected, processed, and stored in bags as blood product units available for blood transfusion.
  A standard autologous leukoreduced packed red blood cell unit will be collected and stored in AS-3 solution in the Columbia University Medical Center blood bank.
  The number of weeks in storage are as follows:
  * 1 week
  * 2 weeks
  * 3 weeks
  * 4 weeks
  * 5 weeks
  * 6 weeks
- Transfusion of PRBC Stored for 6 Weeks: Subjects will receive blood transfusion with packed red blood cells stored for 6 weeks.
  Blood Transfusion: A routine medical procedure in which blood is given through an intravenous (IV) line a blood vessel.
  Packed red blood cells: Red blood cells that have been collected, processed, and stored in bags as blood product units available for blood transfusion.
  A standard autologous leukoreduced packed red blood cell unit will be collected and stored in AS-3 solution in the Columbia University Medical Center blood bank.
  The number of weeks in storage are as follows:
  * 1 week
  * 2 weeks
  * 3 weeks
  * 4 weeks
  * 5 weeks
  * 6 weeks
Period: Overall Study
Arm/Group | Transfusion of PRBC Stored for 1 Week | Transfusion of PRBC Stored for 2 Weeks | Transfusion of PRBC Stored for 3 Weeks | Transfusion of PRBC Stored for 4 Weeks | Transfusion of PRBC Stored for 5 Weeks | Transfusion of PRBC Stored for 6 Weeks
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 8 | 10 | 7 | 8 | 10 | 9
Not Completed | 2 | 0 | 3 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 52 out of the 60 enrolled subjects completed the study and were included in data analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Transfusion of PRBC Stored for 1 Week | Transfusion of PRBC Stored for 2 Weeks | Transfusion of PRBC Stored for 3 Weeks | Transfusion of PRBC Stored for 4 Weeks | Transfusion of PRBC Stored for 5 Weeks | Transfusion of PRBC Stored for 6 Weeks | Total
Number analyzed (Participants) | 8 | 10 | 7 | 8 | 10 | 9 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [23 to 31] | 25 [25 to 31] | 28 [26 to 29] | 28 [25 to 32] | 28 [26 to 33] | 26 [25 to 43] | 27 [25 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 3 | 4 | 3 | 20
  Male | 6 | 6 | 3 | 5 | 6 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 3 | 1 | 1 | 11
  Not Hispanic or Latino | 6 | 7 | 6 | 5 | 9 | 8 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 4 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 1 | 0 | 1 | 5
  White | 6 | 7 | 4 | 5 | 5 | 5 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 7 | 8 | 10 | 9 | 52

OUTCOME MEASURES:

1. Primary Outcome: Non-transferrin-bound Iron Level (AUC)
Description: Area under the curve of change of Non-transferrin-bound iron from immediately after transfusion to end of observation (i.e., from 0-hr after transfusion to 24-hr after transfusion).
Time Frame: 0, 2, 4, 6, 8, 10, 12, 14 and 24 after transfusion
Population: 52 out of the 60 enrolled subjects completed the study and were included in data analysis.
Measure: Median (Inter-Quartile Range); unit: microMole*hr/L
Arm/Group | Transfusion of PRBC Stored for 1 Week | Transfusion of PRBC Stored for 2 Weeks | Transfusion of PRBC Stored for 3 Weeks | Transfusion of PRBC Stored for 4 Weeks | Transfusion of PRBC Stored for 5 Weeks | Transfusion of PRBC Stored for 6 Weeks
Number analyzed (Participants) | 8 | 10 | 7 | 8 | 10 | 9
microMole*hr/L | 0.5588 [-4.153 to 2.959] | 2.839 [-0.02188 to 6.852] | 3.684 [3.509 to 6.864] | 5.272 [0.5483 to 7.754] | 6.416 [4.114 to 9.895] | 39.24 [15.47 to 47.73]

ADVERSE EVENTS:
Time Frame: Up to 24 hours post-transfusion.
Arm/Group | Transfusion of PRBC Stored for 1 Week | Transfusion of PRBC Stored for 2 Weeks | Transfusion of PRBC Stored for 3 Weeks | Transfusion of PRBC Stored for 4 Weeks | Transfusion of PRBC Stored for 5 Weeks | Transfusion of PRBC Stored for 6 Weeks
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/7 | 0/8 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/7 | 0/8 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/7 | 0/8 | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No